CLINICAL TRIAL: NCT04095780
Title: The Effectiveness of Oral Health Promotion on Pneumonia Complicating Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Ya Zhang, Principal Investigator, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81701036
Record Dates: First submitted 2018-10-27; First posted 2019-09-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Pneumonia; Oral Hygiene
Keywords: Oral opportunistic pathogens; Oral health promotion; Pneumonia complicating stroke; Metagenome
MeSH Terms: conditions — Stroke; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced oral hygiene care programme (Experimental): Patients with stroke will receive the advanced oral hygiene care programme (AOHCP) comprising powered tooth brushing and mouth rinsing with chlorhexidine (with a supply of standardized power tooth brushes, mouth rinse, tooth paste and oral hygiene instruction).
  Interventions: Other: Advanced oral hygiene care programme
- Oral hygiene instruction (Experimental): Patients with stroke will only receive the oral hygiene instruction.
  Interventions: Other: Oral hygiene instruction

INTERVENTIONS:
Other: Advanced oral hygiene care programme — 1. Brush teeth with standardized power tooth brush twice a day.
  2. Rinse mouth with chlorhexidine twice a day.
  3. Oral hygiene education
  Arms: Advanced oral hygiene care programme
Other: Oral hygiene instruction — Oral hygiene education
  Arms: Oral hygiene instruction

SUMMARY:
To investigate the evidence for the integration of oral health promotion as part of interdisciplinary stroke rehabilitation.

DETAILED DESCRIPTION:
Pneumonia complicating stroke is very difficult to manage and has a very poor prognosis, leading to a significantly higher risk of death. Oral opportunistic pathogens have been reported to be associated with the incidence of pneumonia among non-stroke immunocompromised subjects. Preliminary studies found that patients with stroke had higher carriage rates of oral opportunistic pathogens than healthy subjects. Therefore, investigators hypothesize that pneumonia complicating stroke is associated with oral opportunistic pathogens, and oral health promotion interventions may reduce the incidence of pneumonia complicating stroke via its effects on the species and relative abundance of oral opportunistic pathogens. In order to prove this, investigators need to (1) firstly conduct a randomized controlled trial to confirm whether oral health promotion is able to reduce the levels of plaque, and the incidence of pneumonia complicating stroke at clinical level; (2) secondly employ metagenomics analysis to compare oral rinse samples and respiratory samples, and to identify pneumonia-associated "oral opportunistic pathogens group"; (3) finally elucidate how oral health promotion influences the species and relative abundance of oral opportunistic pathogens. This proposed study will provide evidence for the integration of oral health promotion as part of interdisciplinary stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* having onset of stroke within 3 days and free of any post-stroke complication
* having moderate to severe functional disability- Barthel Index (BI) scores of <70
* being conscious and respiring voluntarily without ventilator
* not having any lung disease and lower respiratory infection
* not have an indwelling naso-gastric feeding tubes
* having dysphagia as showed by GUSS test (The Gugging Swallowing Screen, GUSS)
* having normal cognitive ability or mild impairment- Mini Mental State Examination (MMSE) >18
* having ability to follow instruction (as an assessment of compliance of oral health intervention)
* not having systemic administration of antibiotics
* not being edentulous

Exclusion Criteria:

* mild disability (Barthel Index > 70)
* having normal swallowing function
* edentulous
* having an indwelling naso-gastric feeding tubes
* having communication disorders, unable to cooperate with family caregivers for oral health promotion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of pneumonia complicating stroke | 1 week
  To calculate and compare the incidence of pneumonia between interventional group and control group, to identify whether the intervention approach could reduce the short-term incidence after the baseline.

SECONDARY OUTCOMES:
The prevalence of pneumonia complicating stroke | 1 month, 3 months, 6 months
  To calculate and compare the long-term incidence of pneumonia between interventional group and control group.
Metagenomic | 3 days, 5 days, 7 days, and 1 month, 3 months, 6 months
  To analyze composition and relative abundance of oral microbiome in oral rinse samples.
Plaque Index | 1 month, 3 months, 6 months
  0 = no plaque detected with probe; 1 = plaque not visible by unaided eye but detectable with probe; 2 = moderate amount of plaque; 3 = abundance of plaque
Gingival Bleeding Index | 1 month, 3 months, 6 months
  0 = no bleeding after probing; 1 = presence of bleeding within 10 seconds after probing.
the Short Form Health Survey 12 (SF-12) | 1 month, 3 months, 6 months
  The SF-12 consists of 12 items covering eight conceptual domains of health: general health (GH), physical functioning (PF), bodily pain (BP), role-physical (RP), mental health (MH), vitality (VT), social functioning (SF), and role-emotional (RE). Four items are reversed for scoring (item no.: 1, 8, 9, and 10). The SF-12 consists of 12 items and each of them has its own physical component summary (PCS) and mental component summary (MCS) regression coefficients. The response to each item will be multiplied by its PCS regression coefficient and added together with the PCS constant to provide Physical Health summary scores (SF-12 PCS). Mental Health summary scores (SF-12 MCS) will be calculated likewise. A higher scores mean a better outcome.
the Oral Health Impact Profile 14 (OHIP-14) | 1 month, 3 months, 6 months
  0=never, 1=hardly ever, 2=occasionally, 3=fairly often, and 4=very often/all of the time. Summary OHIP-14 score and domain scores will be derived by summating responses to each item (i.e. score 2, 3, and 4). A higher scores mean a worse outcome.
the Geriatric Oral Health Assessment Index (GOHAI) | 1 month, 3 months, 6 months
  1 = always, 2 = often, 3 = sometimes, 4 = seldom, and 5= never. Summary GOHAI scores will be derived by summating responses to items after reversing the coding of the three positively worded items (swallowing, appearance, and discomfort when eating). A higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ruoxi Dai, PhD, Study Director — Lecturer
Locations (1):
- The Second People's Hospital of Hefei, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu J, Dai Y, Lo ECM, Qi Y, Zhang Y, Li QL, Dai R. Using metagenomic analysis to assess the effectiveness of oral health promotion interventions in reducing risk for pneumonia among patients with stroke in acute phase: study protocol for a randomized controlled trial. Trials. 2020 Jul 10;21(1):634. doi: 10.1186/s13063-020-04528-3. PMID 32650814